CLINICAL TRIAL: NCT06380946
Title: Influence of Injectable Platelet Rich Fibrin on Different Orthodontic Tooth Movements During Clear Aligner Therapy: A Prospective Clinical Investigation
Brief Title: Influence of Injectable Platelet Rich Fibrin on Different Orthodontic Tooth Movements During Clear Aligner Therapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, farouk ahmed hussein, prinicpaI Investigator, Al-Azhar University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 978/91
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Effect of Platelet Rich FibrinDuring Clear Aligner Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Experimental:iPRF group closure of premolar extraction space (Experimental): closure ofpremolar extraction space that will be performed with iPRFapplication according to a standardized protocol
  Interventions: Biological: iPRF
- intervention group (No Intervention): iPRFgroup closure of premolar extraction space control side
- Experimental: iPRFgroup: distalization intervntion side (Experimental): distalization will be commenced with application of iPRF according to a standardized protocol
  Interventions: Biological: iPRF
- No Intervention: iPRF group: distalization control side (No Intervention): distalization will be commenced without application of iPRF according to a standardized protocol
- Experimental: iPRF group: leveling and alignment (Experimental): leveling and alignment be commenced with application of iPRF according to a standardized protocol
  Interventions: Biological: iPRF
- No Intervention: leveling and alignment without intervention (No Intervention): leveling and alignment without intervention
- Experimental: iPRF group: Intrusion (Experimental): intrusion assisted with application of iPRF according to a standardized protocol
  Interventions: Biological: iPRF
- No Intervention: intrusion control group (No Intervention): intrusion without intervention

INTERVENTIONS:
Biological: iPRF — iPRF has been found to speed up OTM by stimulating the RANK/RANKL/OPG system to initiate osteoclast formation.
  Other Names: injectaleplatelets rich fibrin
  Arms: Experimental: iPRF group: Intrusion; Experimental: iPRF group: leveling and alignment; Experimental: iPRFgroup: distalization intervntion side; Experimental:iPRF group closure of premolar extraction space

SUMMARY:
The aim of this prospective clinical project will be to assess the effect of platelet rich fibrin on the rate of different orthodontic tooth movements during clear aligner therapy.

DETAILED DESCRIPTION:
The aim of this prospective clinical project will be to assess the effect of platelet rich fibrin on the rate of different orthodontic tooth movements during clear aligner therapy.specifically canine retraction,incisors leveling and alignment,maxillary molar distalization and incisors intrusion

ELIGIBILITY:
Inclusion Criteria:A- leveling and alignment Eligibility criteria

1. Age ranges from 15 to 22 years. 2. Bilateral Class II molar relationship. 3. Skeletal Class I or mild Class II relationship. 4. Normal or decreased vertical height. 5. No posterior crowding or spaces. 6. Fully erupted maxillary first and second molars. 7. Congenitally missing or extracted third molars. 8. Good oral hygiene. 9. Absence of any periodontal disease and alveolar bone loss. 10. Absence of medications that may inhibit orthodontic movement

Lower incisor leveling and alignment Inclusion criteria Complete permanent dentition (third molars not included); Moderate mandibular anterior crowding (with little's irregularity index score greater than 4 mm) who required non-extraction approach in the mandibular arch; No tooth size, shape or root abnormalities visible on the patient's radiographic records; No spaces in the mandibular arch; No blocked out tooth that did not allow for placement of the bracket at the

initial bonding appointment; 6. No required management with interproximal stripping, inter-maxillary elastics, open NiTi springs, and removable or extra-oral devices. Canine retraction Eligibility criteria

Age, 15 to 25 years; Class ii division 1 malocclusion with mild or no crowding; No previous orthodontic treatment; No systemic disease that might have affected bone formation or density, such as osteoporosis, hyperparathyroidism, or vitamin d deficiency; Adequate oral hygiene; Probing depth values not exceeding 3 mm across the Entire dentition; Adequate thickness of the attached gingiva (1-2 mm); No radiographic evidence of bone loss

Exclusion Criteria:Patients who required surgery to correct skeletal discrepancies. Patients with congenital dentoskeletal disorders. Missed or mutilated teeth in maxillary arch. Patients with poor oral hygiene and/or periodontally compromised patients Severe dental crowding that necessitates an extraction approach 2. Abnormal anteroposterior and vertical relationships; 3. Patients with cleft lip and palate, anomalies, and syndromes; 4. Previous orthodontic 5. Treatment; 6. Regular medications intake that could interfere with otm. -

-

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Influence of injectable platelet rich fibrin rate of different orthodontic tooth movements by millimeter | post interventionalal at 6months
  rate of orthodontic tooth movement by millimeter

CONTACTS AND LOCATIONS:
Locations (1):
- AlAzhar university, Cairo, Egypt